CLINICAL TRIAL: NCT06739850
Title: Identification of Risk Phenotypes for Sarcopenia Using DXA Whole Body Composition, Anthropometric and Muskuloskeltal Analysis Among Young Adults
Brief Title: Identification of Risk Phenotypes for Sarcopenia Using DXA WBC, Anthropometric and MA Among Young Adults
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHS/Batch-Fall22/002
Record Dates: First submitted 2024-12-14; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group
  Interventions: Combination Product: Identification of Risk Phenotypes of Sarcopenia

INTERVENTIONS:
Combination Product: Identification of Risk Phenotypes of Sarcopenia — Sarcopenia is a condition characterized by progressive loss of skeletal muscle mass, strength, and function, often associated with aging. Traditionally, it is studied in older populations, but your focus is on identifying its early manifestations in young adults, potentially offering a window for prevention.

SUMMARY:
This cross-sectional study aims to identify risk phenotypes for sarcopenia among young adults using Dual-energy X-ray Absorptiometry (DXA) for whole-body composition analysis, along with anthropometric and musculoskeletal assessments. Sarcopenia, characterized by the loss of muscle mass and strength, is a growing concern, particularly among the aging population.

DETAILED DESCRIPTION:
However, early identification in young adults can allow for preventive strategies to improve long-term health outcomes. This study, involving 221 participants aged 15 to 35, focuses on assessing the correlation between DXA-derived body composition, musculoskeletal fitness, and anthropometric measurements with sarcopenia risk. Primary outcome measures include DXA imaging and dynamometry for body composition and strength evaluation, while secondary outcomes focus on detailed anthropometric and musculoskeletal analyses. By addressing early risk factors in younger populations, this research hopes to enhance understanding of sarcopenia's development and support early intervention strategies. Data collection is conducted at the Center of Nuclear Medicine in Lahore, Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* Young Adults ( between 15-35) (7)

Exclusion Criteria:

* Elderly Patients
* Children below the age of 18 Years
* Diagnosed Malignancy
* Diagnosed Patients
* Diseased Individuals such as Chronic Illness and Malignancies

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This cross-sectional study aims to identify risk phenotypes for sarcopenia among young adults using Dual-energy X-ray Absorptiometry (DXA) for whole-body composition analysis, along with anthropometric and musculoskeletal assessments.
Sampling Method: Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
DXA | 12 Months
  DXA Whole Body Imaging is a primary tool of measure for my study

CONTACTS AND LOCATIONS:
Locations (1):
- CENUM Center Mayo Hospital Rd, Anarkali Bazaar, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No